CLINICAL TRIAL: NCT03374046
Title: Apneic Oxygenation in the Pediatric Intensive Care Unit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: K5900309
Record Dates: First submitted 2017-10-24; First posted 2017-12-15 (Actual); Last update posted 2024-10-04 (Actual); Status verified 2024-10

CONDITIONS: Intubation Complication

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Standard care
- Apneic Oxygenation Group (Experimental): During apneic period of intubation attempt, patient will be placed on nasal cannula
  * If 0-2 years: 3L/min NC of 100% FiO2
  * If > or = to 2 through17 years: 5L/min NC of 100% FiO2
  Interventions: Procedure: Apneic Oxygenation

INTERVENTIONS:
Procedure: Apneic Oxygenation — Supplemental oxygen will be provided via nasal cannula during intubation attempt
  Arms: Apneic Oxygenation Group

SUMMARY:
The purpose of the study is to determine the impact of apneic oxygenation on the time to desaturation in pediatric patients treated in a pediatric intensive care unit (PICU). The investigators hypothesize pediatric patients will have an increase in time to desaturation with apneic oxygenation when compared to standard practice in the PICU.

DETAILED DESCRIPTION:
Oxygen (O2) desaturation is one of the risks of intubation, especially in critically ill children with comorbidities, increased O2 consumption and decreased O2 delivery. Desaturation places patients at greater risk for dysrhythmia, hemodynamic instability, hypoxic brain injury, and death. As shown in the oxyhemoglobin dissociation curve, once oxyhemoglobin (PaO2) saturations drop to ~ 90%, there is an increased risk for precipitous desaturation.

Although many may believe there would be no gas exchange during apnea, alveoli continue to take up oxygen even without diaphragmatic movements or lung expansion. As such, the administration of oxygen during intubation (when a patient is apneic) has not been a standard practice until recently.

Recent studies in adults have shown an increase in the time to desaturation when they are given concurrent oxygen administration during an intubation attempt. This use of oxygen during intubation is referred to as apneic oxygenation.

As a result of this work, apneic oxygenation has become standard practice in many emergency departments, even with pediatric patients. Yet, in pediatric hospital units, including intensive care, this is not the standard practice and no pediatric studies have been published on this subject to date.

In the study unit apneic oxygenation is not standard during intubation. The investigators would like to evaluate its use as it has shown benefits in prior research published on adults. Most patients in the PICU are already on a source of oxygen administration prior to intubation, this source of oxygen is usually removed during the intubation attempt, when the patient is apneic and not breathing on his/her own.

Continuing oxygen administration during the apneic period, would be a minimal to no risk intervention and has only shown a benefit during the apneic period.

For this protocol:

Once a decision is made for intubation, the subject will be randomized into one of two groups:

1. Control (standard practice)
2. Apneic oxygenation.

Randomization: Subjects will be stratified by age (0 - 2 years and >2 - 17), randomized in blocks of 10 until the final sample size is achieved.

For all subjects, the study protocol will determine only the provision of supplemental oxygen during intubation.

Decisions regarding the intubation approach, pre-oxygenation, patient positioning, medications used, ventilation strategy, and choice of equipment will be made by the clinical team.

Because of the nature of the study intervention, clinicians and study personnel will be aware of study group assignments after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Treated in the PICU at ACH-PR
* Age 0 through17 years
* Indication for emergent intubation
* Premedication with a paralytic agent resulting in apnea

Exclusion Criteria:

* No paralytic agent used
* Elective intubations
* Presence of cyanotic heart disease
* Inability to safely place nasal cannula on patient
* Nasal intubation
* Patients already enrolled in the study (prior intubation)
* Inability to randomize due to urgency of intubation
* Females who are known to be pregnant

Ages: 0 Days to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 41 (Actual)
Dates: Start 2017-12-23 (Actual); Primary Completion 2020-02-01 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
Time to desaturation | Only during intubation
  To evaluate the effect of apneic oxygenation in time to desaturation (>/= 5% points from baseline O2 saturation) from the onset of apnea during intubation attempts in the PICU

SECONDARY OUTCOMES:
Number of Intubation Attempts | Only during intubation
  To compare the number of intubation attempts prior to successful intubation between children treated with apneic oxygenation compared to standard care

CONTACTS AND LOCATIONS:
Overall Officials: Fasiha Saeed, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Advocate Lutheran General Hospital, Park Ridge, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Weingart SD, Levitan RM. Preoxygenation and prevention of desaturation during emergency airway management. Ann Emerg Med. 2012 Mar;59(3):165-75.e1. doi: 10.1016/j.annemergmed.2011.10.002. Epub 2011 Nov 3. PMID 22050948
- [Background] Taha SK, Siddik-Sayyid SM, El-Khatib MF, Dagher CM, Hakki MA, Baraka AS. Nasopharyngeal oxygen insufflation following pre-oxygenation using the four deep breath technique. Anaesthesia. 2006 May;61(5):427-30. doi: 10.1111/j.1365-2044.2006.04610.x. PMID 16674614
- [Background] Wimalasena Y, Burns B, Reid C, Ware S, Habig K. Apneic oxygenation was associated with decreased desaturation rates during rapid sequence intubation by an Australian helicopter emergency medicine service. Ann Emerg Med. 2015 Apr;65(4):371-6. doi: 10.1016/j.annemergmed.2014.11.014. Epub 2014 Dec 20. PMID 25536868
- [Background] Ramachandran SK, Cosnowski A, Shanks A, Turner CR. Apneic oxygenation during prolonged laryngoscopy in obese patients: a randomized, controlled trial of nasal oxygen administration. J Clin Anesth. 2010 May;22(3):164-8. doi: 10.1016/j.jclinane.2009.05.006. PMID 20400000